CLINICAL TRIAL: NCT03848169
Title: Pulsed Radiofrequency As A Treatment For Mastecatory Muscle Pain In Temporomandibular Disorder Patients
Brief Title: TMD Pulsed Radiofrequency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, JF Asenjo, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-3716
Record Dates: First submitted 2018-08-20; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Temporomandibular Joint Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Ultrasound guidance will be used with a high- frequency linear transducer.After the joint has been identified, the researcher will ask the patient to hold mouth in a neutral position. Masseter, temporalis, medial and lateral pterygoid muscles will be then identified, and with a sterile marker the operator will determine the best point of entry for each muscle injection. Lidocaine 1% will be injected for the skin, always under ultrasound vision. RF needle (18 G, 50 mm of length and active tip of 3 mm) will be inserted into each one of the muscles mentioned previously. Then, through the RF needle, 0.5 ml of normal saline will be injected (to decrease the impedance of the tissues), the electrode will be inserted, and extra-articular PRF will be performed during 4 minutes at 42 degrees Celsius for each muscle. At the end of each muscle treatment, 1 ml of local anesthetic (lidocaine 1%) will be injected through the RF needle, and the needle will be removed.
  Interventions: Other: Radiofrequency
- Control Group (Sham Comparator): Ultrasound guidance will be used with a high- frequency linear transducer. After the joint has been identified, the researcher will ask the patient to hold his or her mouth in a neutral position. Masseter, temporalis and lateral pterigoid muscles will be then identified, and with a sterile marker the operator will determine the best point of entry for each muscle injection (mainly over the most common sites of trigger points for the masticatory muscles). Lidocaine 1% will be injected for the skin, always under ultrasound vision. RF needle (18 G, 50 mm of length and active tip of 3 mm) will be inserted into each one of the muscles mentioned previously. Then, through the RF needle, an electrode will not be inserted, but a simulation for PRF will be done during 4 minutes for each muscle (sham). At the end of each muscle puncture, 1 ml of local anesthetic (lidocaine 1%) will be injected through the needle, and the needle will be removed.
  Interventions: Other: Radiofrequency

INTERVENTIONS:
Other: Radiofrequency — See previous page

SUMMARY:
PRF of the masticatory muscles (masseter, temporalis, medial and lateral pterygoid muscle) can improve pain intensity and functional recovery of the jaw in patients with extra-articular TMD.

DETAILED DESCRIPTION:
The temporomandibular joint is formed by the mandibular condyle inserting into the mandibular fossa of the temporal bone. Muscles of mastication are primarily responsible for the movement of this joint. Its functionality may be affected by different disorders that are characterized by craniofacial pain involving the joint, masticatory muscles, or muscle innervations of the head and neck. These are known as temporomandibular disorders (TMD). It affects 10% to 15% of adults, but only 5% seek treatment. The incidence of TMD peaks from 20 to 50 years of age and are more common in female population.

TMD is categorized as intra-articular (within the joint) or extra-articular (involving the surrounding musculature). Musculoskeletal conditions (myofascial pain disorder) are the most frequent cause of TMD, accounting for at least 50% of cases. Thus, musculoskeletal conditions associated with TMD include spasm and/or tenderness to palpation of the masseter, temporalis, and/or pterygoid muscles.

Etiology of TMD is multifactorial. Factors consistently associated with TMD include other pain conditions, fibromyalgia, autoimmune disorders, sleep apnea and psychiatric illness. According to the literature, there is 1.8-fold increase in myofascial pain in people with anxiety.

It is important to mention that patients with TMD present with an increase risk to develop chronic and intense headaches. The relationship between chronic TMD and various headaches could be due to similarity in the pathophysiology of both diseases.4-6 Studies suggest, that the trigeminal nucleus contribute to central sensitization associated to interference in descending modulation, and could produce the amplification of pain in this region.

Treatment for TMD is complicated and requires specific knowledge and exercises to strengthen some groups of muscles and stretch others, occlusal splint therapy, massage, trigger point injections, and pharmacotherapy. Although the management seems difficult, most of the patients experience successful improvement once a proper protocol has been established. Muscle relaxants (baclofen, tizanidin, cyclobenzaprine), nonsteroidal anti-inflammatory drugs (NSAIDS), opioids, anticonvulsants (e.g., gabapentin), ketamine, tricyclic antidepressants (e.g., amitriptyline) and benzodiazepines, have also been used clinically for TMD management, but there is no evidence that supports or refutes the effectiveness of these medications. In some cases where patients present with severe acute pain, or chronic pain secondary to serious TMD, inflammation, or degeneration, minimally invasive and invasive procedures should be considered.

As a general concept, pain treatment by radiofrequency (RF) energy is a technique widely used in the pain practice. RF denervation is a percutaneous procedure involving the destruction of nerves using heat generated by a RF current. The basic principles of RF, involve transferring an alternating electrical current by a generator to a nerve via an active electrode. The electrode is introduced through an insulated needle, with the exposed active tip transferring the current to the surrounding tissues.

It is worth mentioning that for interventional pain management purposes there are different modes of RF that could be used: the continuous RF (CRF) lesion where the heat generated causes tissue coagulation over 65 degrees Celsius, and the pulsed RF (PRF), which is a non-destructive procedure where electrical bursts of 20 milliseconds of electricity are applied followed by 480 milliseconds of no current to allow heat to dissipate, keeping the tissue temperature below 42 degrees Celsius. Even though different theories have been suggested for PRF mechanism of action, Vallejo et al. propose that PRF is able to modulate nerve electrical conduction, and the therapeutic effect is the result of the electrical field, where c-fos activation and potential effect over the norepinephrine and serotonin systems have been involved.

Several studies point to a thermal physical effect of PRF for myofascial pain syndrome. It is proposed, that PRF acts delivering the electric field and heat bursts to the targeted tissues, without damaging these structures, and blocking the central sensitization and producing a better response of the downward pathways of pain. So far, several studies have reported the positive effect of PRF on managing pain syndrome mainly for trapezius muscle and gastrocnemius.

Tamimi et al, published a case series of PRF treatment for myofascial trigger points and scar neuromas. They found that 89% of the patients with longstanding myofascial or neuromatous pain that was refractory to previous treatments, experienced 75-100% reduction in their pain following PRF management. The researchers also found that 67% of the patients experienced 6 months to greater than one year of pain relief. Despite the small size of the sample, the authors conclude that PRF could be a minimally invasive, less neurodestructive treatment modality for these painful conditions.

Taking in consideration previous facts mentioned above and the lack of strong and high-quality evidence for the use of PRF for extra-articular TMD, there is a specific interest to develop a prospective pilot study to test the application of this technique into the main affected muscles that contribute for development of temporomandibular pain. PRF could be an alternative that might offer an effective way to treat pain in this population with myofascial origin of pain. Hence, the purpose of this research is to evaluate the improvement of temporomandibular pain intensity and functionality of the jaw, after extra-articular PRF in patients with TMD.

ELIGIBILITY:
Inclusion Criteria:

* Thirty consecutive patients, male and female, between 18 and 80 years old, with extra-articular TMD as diagnosed by a specialist of the Maxillofacial team based on Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD) for Clinical and Research Applications, with chronic pain related to TMD (for more than three months according to IASP definition), and who have plateaued with conventional treatment in the past three months, will be prospectively recruited at the Maxillofacial Surgery Clinic

Exclusion Criteria:

* • Patients younger than 18 years old.

  * ASA physical status >3,
  * Contraindication for local anesthetics or RF.
  * Immunosuppression or high risk of infection.
  * Coagulation impairment.
  * Patients with psychiatric illness.
  * Patients with cognitive impairment.
  * Patients currently taking opioids.
  * Patients that had botulinum toxin or steroid injections in the head or neck area in the past three months.
  * Patient with pacemaker.
  * Patient with prosthetic joint replacement, or placement of any metallic surgical device in or around the area of treatment.
  * Infection of the TMJ.
  * Muscular dystrophy.
  * Pathology or impaired masticatory muscles.
  * Pregnancy.
  * Autoimmune diseases.
  * Arthralgia or intra-articular joint dysfunction.
  * Patients with allergy to Cefazolin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in static and dynamic TMD pain | 30 minutes, 4 and 12 weeks post procedure
  using Numerical Rating Scale (NRS) at the end of the procedure (NRS post-procedure), and in the follow-up at 4 weeks and 12 weeks post-procedure.

SECONDARY OUTCOMES:
change in maximal mouth opening | 30 minutes, 4 and 12 weeks post procedure
  by measurement of maximum mouth opening (MMO) in centimetres
Pain medications use | 30 minutes, 4 and 12 weeks post procedure
  In oral morphine equivalence
Change in lateral jaw excursion | 30 minutes, 4 and 12 weeks post procedure
  By measurement of lateral jaw excursion in centimetres
Change in jaw protrusion | 30 minutes, 4 and 12 weeks post procedure
  By measurement of jaw protrusion in centimetres

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided